CLINICAL TRIAL: NCT07170111
Title: Predictive Factors for the Success of Greater Occipital Nerve Block in Migraine: A Multicenter Prospective Study
Brief Title: Predictors of GON Blockade Success in Migraine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Collaborators: Umraniye Education and Research Hospital (Other Government); Gaziantep City Hospital (Other); Namik Kemal University School of Medicine, Tekirdag (Other); Bakırçay University, Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, Tuba Tanyel Saraçoğlu, Medical Doctor, Başakşehir Çam & Sakura City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25.06.2025.242
Record Dates: First submitted 2025-08-22; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Migraine
Keywords: migraine; GON block; greater occipital nerve; greater occipital nerve block; predictive factors
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GON Block Group (Experimental)
  Interventions: Procedure: Greater Occipital Nerve (GON) Blockade

INTERVENTIONS:
Procedure: Greater Occipital Nerve (GON) Blockade — The greater occipital nerve block (GONB) will be performed using anatomical landmarks (distal approach). The injection point is located at the medial one-third of the line between the external occipital protuberance and the mastoid process. A 26-gauge insulin needle will be used for the procedure. The block will be administered bilaterally with 0.5% bupivacaine, 1.5 ml per side (total 3 ml). The intervention will be repeated once weekly for a total of four sessions

SUMMARY:
This multicenter, prospective cohort study aims to identify clinical and demographic predictors that influence the success of greater occipital nerve (GON) block in patients with migraine.

Patients will be evaluated at baseline, on each injection day, and at one- and three-month follow-ups. Study parameters include demographics, migraine type and duration, comorbidities, headache characteristics, treatment history, and validated outcome measures such as the Numeric Rating Scale (NRS), Headache Impact Test-6 (HIT-6), and Global Rating of Change (GRoC).

The goal is to establish predictive factors of treatment success in order to optimize patient selection and contribute robust multicenter evidence to individualized migraine management

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine for at least 6 months, according to ICHD-3 criteria
* Age between 18 and 65 years
* Inadequate response to preventive therapy used regularly for at least 3 months
* Planned treatment with greater occipital nerve block (GONB) and provision of signed informed consent
* Receiving GONB treatment for the first time

Exclusion Criteria:

* Pregnancy or breastfeeding
* Presence of malignancy
* Coagulopathy or anticoagulant therapy
* Local infection, open wound, or history of surgery at the injection site preventing the procedure
* History of severe neurological or psychiatric disorders
* Receipt of interventional treatment (e.g., Botox, acupuncture, neural therapy, nerve blocks) within the last 3 months
* Use of steroids or immunosuppressive therapy
* Start of a new preventive therapy within the last 3 months
* Inability to comply with keeping a headache diary
* Known hypersensitivity or allergy to bupivacaine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of days with headache | Baseline,1st month and 3rd month

SECONDARY OUTCOMES:
The 6-Item Headache Impact Test (HIT-6) | Baseline,1st month and 3rd month
  The 6-Item Headache Impact Test (HIT-6) is a brief, validated questionnaire that assesses the adverse impact of headaches on daily functioning, with higher scores indicating greater impact.
Global Rating of Change (GROC) | 1st month and 3rd month
  The Global Rating of Change (GROC) is a patient-reported scale that measures perceived change in health status over time, typically ranging from very much worse to very much improved.
Numeric Rating Scale | Baseline,1st month and 3rd month
  A simple and widely used tool to assess pain intensity, where patients rate their pain on a scale from 0 to 10, with 0 meaning 'no pain' and 10 meaning 'the worst pain imaginable
Number of migraine attacks | Baseline, 1st month and 3rd month
Duration of migraine attacks | Baseline, 1st month and 3rd month
Analgesic consumption | Baseline, 1st month and 3rd month

CONTACTS AND LOCATIONS:
Locations (1):
- Başakşehir Çam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No